CLINICAL TRIAL: NCT00741052
Title: Randomized, Double Blind, Controlled Clinical Trial to Evaluate the Efficacy of Multiple-dose Ciprofloxacin With Single Dose Azithromycin Therapy for Adults With Cholera Due to Multiply Resistant Strains of V. Cholerae O1 or O139
Brief Title: Ciprofloxacin Multiple Dose for Adult Cholera
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Diseases Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-022
Record Dates: First submitted 2008-08-04; First posted 2008-08-26 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2008-08

CONDITIONS: Cholera
Keywords: V. cholerae,; ciprofloxacin,; azithromycin,; randomized
MeSH Terms: conditions — Cholera | interventions — Ciprofloxacin; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ciprofloxacin
  Interventions: Drug: Ciprofloxacin
- 2 (Active Comparator): Azithromycin
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Ciprofloxacin — 12 hourly oral dose of ciprofloxacin for 3 days
  Other Names: BEOFLOX
  Arms: 1
Drug: Azithromycin — 1 gm Azithromycin single dose
  Other Names: TRIDOSIL
  Arms: 2

SUMMARY:
Cholera is an important diarrhoeal disease and an important cause of death, particularly during epidemic outbreaks, in Bangladesh and many other developing countries. Used as an adjunct to management of dehydration, antimicrobial therapy using an appropriate agent reduces diarrhoea duration and stool volume in severe cholera by about half.

The usefulness of antimicrobials has, however, been greatly eroded by the increasing prevalence of resistant strains of V. cholerae O1. From October 2004 at the Matlab Hospital and from December 2004 at the Dhaka Hospital of ICDDR, B, V. cholerae strains became increasingly resistant to tetracycline and erythromycin- two drugs used in the treatment of severe cholera in adults and children respectively. Because of this high prevalence of resistance we resorted in early 2005 to using ciprofloxacin for treatment against multi drug resistant V. cholerae. Although all isolates were susceptible to ciprofloxacin when standard thresholds for disc-diffusion or E-test were used, but majority of the strains demonstrated a MIC value of 0.250 µg/ml, over hundred-folds greater than the V. cholerae strains tested in earlier years, which generally had a MIC of <0.003 µg/ml.

In this randomized, double blind, controlled trial we will assess clinical and bacteriological response to 12 hourly oral dose of ciprofloxacin for 3 days in which the first two doses will be 1 g each and the later 4 doses will be 500 mg each, and compare them with a single 1 g oral dose of azithromycin. We are using azithromycin as the comparator drug because current circulating V. cholerae isolates are susceptible (MIC ≤ 0.125 µg/ml) to this azithromycin, and single-dose azithromycin has been evaluated earlier to be effective in the treatment of cholera.

DETAILED DESCRIPTION:
Cholera is caused by infection of the human intestine with Vibrio cholerae O1 or V. cholerae O139. It is a major health problem in many developing countries including Bangladesh.1 The importance of cholera as a worldwide public health problem is evident from the large number of countries affected by cholera epidemics.2 Data of the Diarrhoeal Disease Surveillance system of the Dhaka Hospital demonstrated that V. cholera O1 was the most frequently isolated pathogens (617/2,068 i.e. 30%) in patients attending the hospital with diarrhoeal illnesses in 2006. By extrapolating the number of patients enrolled in the surveillance system we estimate that over 30,000 out of the total 106,531 patients attending the hospital in 2006 had cholera- a huge number of patients indeed.

Like other diarrhoeal illnesses, prevention and management of dehydration using appropriate oral and/or intravenous fluids is the mainstay in the management of cholera, irrespective of severity. However, appropriate antimicrobial therapy is a very useful adjunct therapy that reduces the duration of diarrhoea, the volume of diarrhoeal stools (thus the amount of oral and intravenous fluids), and also the duration of faecal excretion of the pathogen, V. cholerae O1 and O139 by about 50%. 3-6 Based on these observations made in numerous clinical trials, routine use of an appropriate antimicrobial therapy is recommended in the management of severe cholera, both in adults and children. All three benefits, as described above, are very important in resources-constraint settings where cholera is endemic and also during epidemic outbreaks.

Nosocomial transmission of cholera has also been increasingly recognized as an important problem,7 and reducing the duration of excretion of Vibrio cholerae in the stool associated with appropriate antimicrobial therapy will presumably decrease the rate of nosocomial infection. Lastly, by shortening the course of illness, patients and their families' can more quickly return to their normal life, lessening their financial burden, which is of particular relevance to socio-economically disadvantaged population who disproportionately share the most of the disease burden from cholera.

From the time of the initial controlled trials of antimicrobial therapy for cholera, almost four decades ago,3 a number of antimicrobial agents have been evaluated to be useful in the treatment of cholera. Tetracycline, chloramphenicol, doxycycline, furazolidone and trimethoprim-sulfamethoxazole have all been found to be effective in the treatment of cholera when given in multiple doses for 3 days.8-14 Tetracycline and it's long-acting congener doxycycline are also effective when administered in a single 1 or 2 g and 200 or 300 mg oral doses respectively in adults.13, 14 Vomiting is a common problem in association with doxycycline therapy and the problem is greater when doxycycline is used in 300 mg dose (39%) compared to when 200 mg dose is used (30%); however, the therapeutic efficacy is better with the higher dose (mean duration of diarrhoea were 32h vs. 40h respectively.14

Antimicrobial resistance has now become an important problem in the clinical management of cholera. For example, in 2006 virtually all of the 683 clinical strains of V. cholerae O1 isolated from patients attending the Dhaka Hospital were multiply drug resistant with 100% resistance to ampicillin, furazolidone and co-trimoxazole, 83% to erythromycin and 85% to tetracycline.15 All V. cholerae strains remained susceptible to ciprofloxacin by disc-diffusion testing, but in E-test their MIC were noted to have increased from 0.002 µg/ml during 1993-2003 to 0.250-0.380 µg/ml in 2006

Resistance of V. cholerae to commonly used drugs such as tetracycline, doxycycline, furazolidone and trimethoprim-sulfamethoxazole have also been reported from Asia, Africa and Latin America,17-20 In the early 1990's increasing prevalence of V. cholerae resistant to antimicrobials commonly used in the treatment of cholera (tetracycline, ampicillin, co-trimoxazole) prompted our group and others to conduct series of trials to identify newer affective agents for treatment of cholera. We evaluated ciprofloxacin in both adult and children infected with V. cholerae O1 and O139, and observed very good rates of both clinical and bacteriological response when used in multiple doses or in a single dose administered only once.11, 21, 22

Ciprofloxacin, is a member of the class of drugs called fluoroquinolones, which act by blocking the action of bacterial DNA gyrase.23 This enzyme, which is not present in human cells, is responsible for supercoiling of bacterial DNA, an essential element for DNA functions.24 Without the three-dimensional DNA structure the cell is unable to replicate, and thus bacterial growth is rapidly halted. Ciprofloxacin is the most active of the fluorinated 4-quinolones (ciprofloxacin, norfloxacin, ofloxacin) against bacterial diarrhoea pathogens in-vitro as assessed by MIC. It has a relatively long serum half-life.25 Due to its multiple mechanisms of excretion toxic levels of quinolones do not usually accumulate in the body. Experience suggests that resistance against ciprofloxacin develops much more slowly than against the older quinolone agent such as nalidixic acid, as the rate of spontaneous mutation is much lower and multiple mutations are required to confer frank resistance.26, 27 Increases in the MIC, however, can occur with single mutation, and this is the likely sequence that has occurred among currently circulating V. cholerae isolates in Bangladesh.

Because of resistance to other agents and susceptibility of the isolates to ciprofloxacin in-vitro, disc diffusion tests, Dhaka and Matlab Hospitals of ICDDR, B changed their treatment policy (early 2005) to single-dose ciprofloxacin therapy for treatment of cholera irrespective of patients' age, except for cholera in pregnant women. However, experienced physicians at the Dhaka Hospital quickly noted sub-optimal clinical response to ciprofloxacin therapy- higher stool output and longer hospitalisation. A quick review of the clinical study that we recently published in the New England Journal of Medicine confirmed these findings.28 In that study only 26 (27%) of 98 patients who were infected with V. cholerae O1 experienced an optimal clinical response to single-dose ciprofloxacin, while only 10 (10%) of the 98 patients had a bacteriologic cure, as defined in the protocol. Eventual determination of MICs of the V. cholerae strains from that study revealed that the inferior clinical and bacteriological response to ciprofloxacin was associated with an increase in MIC values.29 Table 1 below shows the increase in ciprofloxacin MIC values that were observed during 1993-1994 when we first conducted clinical trials with ciprofloxacin to subsequent years including in 2005 when ciprofloxacin was first introduced for routine use in the treatment of cholera at the Dhaka Hospital. We can see, the median MICs has increased approximately one hundred folds between 1993 and 2006.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 60 years.
* Gender: Male
* Duration of diarrhoea: Not exceeding 24 hours
* Written informed consent for participation.
* Dehydration status: Severe dehydration.
* Positive stool dark-field microscopic examination for V. cholerae & culture positive for V cholerae
* For patients assigned to receive ciprofloxacin, an MIC of the V. cholerae isolates to ciprofloxacin of > 0.190 µg/ml and to azithromycin of ≤ 0.125 µg/ml.

Exclusion Criteria:

* History of receiving an antimicrobial agent known to be effective in cholera in adults.
* Concomitant infection requiring antimicrobial therapy other than the study drugs.
* Chronic illness.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine whether clinical success of therapy in the two treatment regimens are comparable. | 48 hours

SECONDARY OUTCOMES:
Compare the rates of bacteriological success. Compare the diarrhea duration. Compare stool volume of patients. Measure stool concentrations of the two drugs and compare them with MICs of V. cholerae. Record and compare adverse events. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wasif A Khan, MBBS, MS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh